CLINICAL TRIAL: NCT06315426
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of GR1802 Injection in Combination With Background Therapy in Patients With SAR.
Brief Title: A Study of IL4Rα Monoclonal Antibody in Patients With Seasonal Allergic Rhinitis(SAR).
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-011
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interleukin-4 receptor responder 1 (Experimental)
  Interventions: Biological: GR1802 injection
- Interleukin-4 receptor responder 2 (Experimental)
  Interventions: Biological: GR1802 injection
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GR1802 injection — Recombinant fully human anti-IL4Rα monoclonal antibody drug.
  Arms: Interleukin-4 receptor responder 1; Interleukin-4 receptor responder 2
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) is a non-infectious chronic inflammatory disease of the nasal mucosa mainly mediated by immunoglobulin E after exposure to allergens in atopic individuals. The typical symptoms of AR are paroxysmal sneezing, watery rhinorrhea, itching, and nasal congestion, which may be accompanied by ocular symptoms, including eye itching, tearing, redness, and burning sensation, which are more common in patients with hay fever allergies. Bronchial asthma is associated with bronchial asthma in 40% of patients with AR, suggesting a comorbid feature of allergic disease.

ELIGIBILITY:
Main Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. Seasonal allergic rhinitis has been prevalent for at least 2 years.
3. Poor control of seasonal allergic rhinitis with nasal glucocorticoids or other therapeutic agents during the same pollen season in the past.
4. Positive SPT or serum-specific IgE test results.
5. Symptom severity scores for the season met the enrollment criteria.

Main Exclusion Criteria:

1. Other nasal comorbidities or co-morbidities/states that may be present at the time of screening that affect efficacy determination.
2. Subjects whose allergen exposures in their home or work environments may be expected to change significantly during the trial period.
3. Subjects with poorly controlled recent asthma conditions.
4. Presence of current or past history of infection of special concern, e.g., active tuberculosis, helminthic infections, severe herpes virus infections, etc.
5. Previous use of anti-interleukin 4 receptor alpha subunit (IL4Rα) monoclonal antibody.
6. Have a serious underlying medical condition that, in the opinion of the investigator, may pose a risk to subject safety by participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-03-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in rTNSS( reflective total nasal symptom scores) | Over 2 weeks
  TNSS is the sum of the four symptom scores of runny nose, nasal congestion, nasal itching, and sneezing, with each symptom scoring from 0 to 3. The total score is 12, the higher the score, the worse the symptoms.

SECONDARY OUTCOMES:
Change from Baseline in rTOSS( reflective total ocular symptom scores) | Over 2、4 weeks
  TOSS is the sum of symptom scores of eye itching/foreign body sensation/redness and tearing, with each symptom scoring from 0 to 3. The total score is 6, the higher the score, the worse the symptoms.
Change from Baseline in rTNSS | Over 4 weeks
  TNSS is the sum of the four symptom scores of runny nose, nasal congestion, nasal itching, and sneezing, with each symptom scoring from 0 to 3. The total score is 12, the higher the score, the worse the symptoms.
Mean change from baseline in iTNSS(instantaneous total nasal symptom scores) | week 2、4
  TNSS is the sum of the four symptom scores of runny nose, nasal congestion, nasal itching, and sneezing, with each symptom scoring from 0 to 3. The total score is 12, the higher the score, the worse the symptoms.
Mean change from baseline in iTOSS(instantaneous total ocular symptom scores) | week 2、4
  TOSS is the sum of symptom scores of eye itching/foreign body sensation/redness and tearing, with each symptom scoring from 0 to 3. The total score is 6, the higher the score, the worse the symptoms.
Change from baseline in VAS(Visual Analog Scale) score | week2、4
  Patients marked the score corresponding to the severity of the current overall AR symptoms by drawing a line on a 0-10 cm scale，the higher the score, the worse the symptoms.
Change from baseline in RQLQ(Rhinoconjunctivitis Quality of Life Questionnaire) scores | week2、4
  The RQLQ is used to measure the problems that adults with rhinoconjunctivitis experience in their daily lives. It has 28 questions in 7 domains. The total score is the sum of the 7 domain scores, with higher scores being associated with poorer quality of life.
Adverse events (AEs) | up to 12 weeks
  Incidence of AEs.
Immunogenicity characteristics | up to 12 weeks
  Positive rate of ADA(anti-drug antibody) testing

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, PHD, Principal Investigator — Tongji Hospital
Locations (15):
- China (15):
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Central Hospital of Qinghe County, Xingtai, Hebei
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan